CLINICAL TRIAL: NCT04529148
Title: Randomized, Double-masking, Placebo-controlled, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Ginkgo Biloba Dropping Pills in the Treatment of Coronary Heart Disease With Stable Angina Pectoris and Depression
Brief Title: The Efficacy and Safety of Ginkgo Biloba Dropping Pills in the Treatment of Coronary Heart Disease With Stable Angina Pectoris and Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Collaborators: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WanbangdePharm
Record Dates: First submitted 2020-08-20; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Stable Angina Pectoris Associated With Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The treatment group (Experimental): Ginkgo biloba dropping pills (63mg / pill), oral, 5 pills each time, three times a day,12 weeks totally. ( Continued to receive the best western medicine treatment for stable angina pectoris of coronary heart disease during the observation period.)
  Interventions: Drug: Ginkgo biloba dropping pills，best western medicine treatment
- The control group (Placebo Comparator): Mimetic drug of ginkgo biloba dropping pills (63mg / pill),oral, 5 pills each time, three times a day,12 weeks totally.( Continued to receive the best western medicine treatment for stable angina pectoris of coronary heart disease during the observation period.)
  Interventions: Drug: Mimetic drug of ginkgo biloba dropping pills，best western medicine treatment

INTERVENTIONS:
Drug: Ginkgo biloba dropping pills，best western medicine treatment — oral
  Arms: The treatment group
Drug: Mimetic drug of ginkgo biloba dropping pills，best western medicine treatment — oral
  Arms: The control group

SUMMARY:
To evaluate the clinical efficacy of Ginkgo biloba dropping pills on improving the frequency of angina pectoris and the life quality of patients with stable angina pectoris and depression symptoms on the basis of the best western medicine treatment; Study on the clinical pharmacological mechanism of Ginkgo biloba dropping pills.

DETAILED DESCRIPTION:
This is a randomized, double-masking, placebo-controlled, multicenter clinical trial. The 72 subjects will be divided into experimental group and control group. The experimental group will be given Ginkgo biloba dropping pills (63mg / pill) , oral, 5 pills each time, three times a day. The control group will be given mimetic drug of ginkgo biloba dropping pills (63mg / pill) , oral, 5 pills each time, three times a day, for 12 weeks to evaluate the effect of Ginkgo biloba dropping pills on coronary heart disease Efficacy and safety of stable angina pectoris with depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years , regardless of gender;
2. Clearly understand and voluntarily participate in the study, and sign the informed consent form;
3. In accordance with the diagnosis of coronary heart disease, and the following diagnostic criteria meet at least one of the following criteria: ① have a clear history of myocardial infarction; ② have accept the treatment of coronary artery revascularization; ③ coronary radiography or coronary angiography results show that at least one coronary artery stenosis and lumen stenosis ≥ 50%; ④ cardiac magnetic resonance imaging or radionuclide myocardial perfusion imaging or cardiac color Doppler diagnosis Coronary heart disease with myocardial ischemia;
4. Consistent with the diagnosis of stable angina pectoris;
5. Stable angina pectoris has been treated according to the clinical guidelines and has been stable for at least 4 weeks;
6. Meet the diagnostic criteria for depressive episode in 《the international statistical classification of diseases and related health problems (ICD-10)》 issued by the World Health Organization;
7. In the past 7 days, have not used any food that has an impact on intestinal flora, such as foods containing probiotics (such as yogurt) or drugs (such as antibiotics).

Exclusion Criteria:

1. Acute myocardial events, unstable angina pectoris, severe heart failure; serious arrhythmia; severe or poorly controlled hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg); sitting blood pressure and systolic blood pressure ≤ 85 MmHg or symptomatic hypotension, severe primary diseases such as liver, kidney and hematopoietic system, or serious diseases affecting their survival (such as tumor, etc.);
2. Serious suicidal tendency; Hamilton Depression Scale item 3 ≥ 3; bipolar disorder depressive episode in patients with epilepsy history, or depression secondary to other mental or physical diseases; alcohol and drug dependence within one year;
3. Abnormal liver and kidney function (ALT and / or AST > 3 times of the upper normal limit, and / or CRE > 2 times of the upper normal limit);
4. Patients who are currently taking anti anxiety drugs;
5. Pregnant women, lactating women, women of childbearing age who do not take effective contraceptive measures, or who plan to conceive during the trial, and whose pregnancy test results are positive before the test;
6. Those who have participated in clinical trials of other new drugs within 30 days before screening;
7. Other reasons the researcher thinks it is not suitable to participate in the experiment;
8. Those with allergic constitution are allergic to the ingredients contained in Ginkgo biloba dropping pills;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-09-20 (Estimated); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Score of Seattle Angina Questionnaire（SAQ ） | at the 0-week
  Score 19 items of the 5 items of the scale, and calculate the total scores of the 5 items respectively, then convert them into standard points according to the formula: standard score = (actual score of the dimension - lowest score of the dimension) / (highest score of the dimension - lowest score of the dimension) × 100. The higher the score, the better the quality of life and body function.
Score of Seattle Angina Questionnaire（SAQ ） | at the 4-week
  Score 19 items of the 5 items of the scale, and calculate the total scores of the 5 items respectively, then convert them into standard points according to the formula: standard score = (actual score of the dimension - lowest score of the dimension) / (highest score of the dimension - lowest score of the dimension) × 100. The higher the score, the better the quality of life and body function.
Score of Seattle Angina Questionnaire（SAQ ） | at the 8-week
  Score 19 items of the 5 items of the scale, and calculate the total scores of the 5 items respectively, then convert them into standard points according to the formula: standard score = (actual score of the dimension - lowest score of the dimension) / (highest score of the dimension - lowest score of the dimension) × 100. The higher the score, the better the quality of life and body function.
Score of Seattle Angina Questionnaire（SAQ ） | at the 12-week
  Score 19 items of the 5 items of the scale, and calculate the total scores of the 5 items respectively, then convert them into standard points according to the formula: standard score = (actual score of the dimension - lowest score of the dimension) / (highest score of the dimension - lowest score of the dimension) × 100. The higher the score, the better the quality of life and body function.
Frequency of angina pectoris related symptoms every week | at the 0-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 1-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 2-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 3-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 4-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 5-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 6-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 7-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 8-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 9-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 10-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 11-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.
Frequency of angina pectoris related symptoms every week | at the 12-week
  With the help of questionnaire survey，we can judge whether there is angina pectoris，record the frequency of angina pectoris symptoms, and the frequency before treatment, during follow-up and after treatment will be compared within and between groups.

SECONDARY OUTCOMES:
The Short Form-36 Health Survey | at the 0-week
  The 35 items of SF-36 quality of life scale were summarized into 8 dimensions. According to the influence degree of each item on the quality of life, the corresponding weight was given, and each dimension was converted into 100 points. The higher the score, the better the functional status and the higher the quality of life.
The Short Form-36 Health Survey | at the 12-week
  The 35 items of SF-36 quality of life scale were summarized into 8 dimensions. According to the influence degree of each item on the quality of life, the corresponding weight was given, and each dimension was converted into 100 points. The higher the score, the better the functional status and the higher the quality of life.
Hamilton Depression Scale (HAMD-17) | at the 0-week
  All items in the 17 items were scored，the scores of minimum values is 0, the maximum values is 52，the higher the score, the more serious the depression，after treatment，the score reduction rate ≥ 50% is defined as valid.
Hamilton Depression Scale (HAMD-17) | at the 12-week
  All items in the 17 items were scored，the scores of minimum values is 0, the maximum values is 52，the higher the score, the more serious the depression，after treatment，the score reduction rate ≥ 50% is defined as valid
Composite endpoint incidence of major adverse cardiovascular events (MACE) | at the 12-week
  Record the major adverse cardiovascular events (MACE)（Mace including cardiovascular death, non fatal myocardial infarction, revascularization）.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Foshan Chancheng Central Hospital, Foshan, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Shenzhen Luohu District People's Hospital, Shenzhen, Guangdong
  - The Second Affiliated Hospital of Guizhou University of Chinese Medicine, Guiyang, Guizhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu T, Li S, Li Z, Long W, Liu Q, Tang H, Huang X, Tang Y, Dong X, Ning Y, Tian S, Xu T, Xian SX, Liao H, Hong Y, Yang Z. Efficacy and safety of Ginkgo biloba dropping pills in the treatment of coronary heart disease with stable angina pectoris and depression: study protocol for a randomised, placebo-controlled, parallel-group, double-blind and multicentre clinical trial. BMJ Open. 2023 May 10;13(5):e055263. doi: 10.1136/bmjopen-2021-055263. PMID 37164472
- [Derived] Tully PJ, Ang SY, Lee EJ, Bendig E, Bauereiss N, Bengel J, Baumeister H. Psychological and pharmacological interventions for depression in patients with coronary artery disease. Cochrane Database Syst Rev. 2021 Dec 15;12(12):CD008012. doi: 10.1002/14651858.CD008012.pub4. PMID 34910821